CLINICAL TRIAL: NCT01808755
Title: Recurrent Urinary Tract Infections in Adult Women: a Pilot Study With Oral D Mannose
Brief Title: D Mannose in Recurrent Urinary Tract Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Daniele Porru, Consultant Urologist, Principal investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DMannose UTIs
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Results first posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-04

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: recurrent urinary tract infections; D Mannose; cystitis; antibiotic treatment
MeSH Terms: conditions — Urinary Tract Infections; Cystitis | interventions — Mannose; Sugars; Trimethoprim, Sulfamethoxazole Drug Combination; Trimethoprim; Sulfamethoxazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D Mannose (Experimental): 1 gr. every 8 hours for 2 weeks, subsequently 1 gr. every 12 hours for 22 weeks
  Interventions: Dietary Supplement: D Mannose; Drug: trimethoprim/sulfamethoxazole
- trimethoprim/sulfamethoxazole (Active Comparator): intervention was a 5-days course of trimethoprim/sulfamethoxazole cp 160 mg/800 mg twice a day. Then one week of antibiotic every 4 weeks for the following 23 weeks
  Interventions: Dietary Supplement: D Mannose; Drug: trimethoprim/sulfamethoxazole

INTERVENTIONS:
Dietary Supplement: D Mannose — 1 gr. every 8 hours
  Other Names: sugar
Drug: trimethoprim/sulfamethoxazole — one cp b.i.d. for 5 days. Then one week of antibiotic every 4 weeks for the following 23 weeks
  Other Names: trimethoprim/sulfamethoxazole 160 mg/800 mg

SUMMARY:
Background- In recurrent urinary tract infections (RUTIs) usual prophylactic antibiotic regimes do not change the long term risk of recurrence.

Objective- D-Mannose is a sugar, it sticks to E. coli bacteria, the aim of the study was to evaluate its efficacy in the treatment and prophylaxis of recurrent UTIs.

Design, setting and participants- : In this crossover trial female patient were eligible for the study if they had recurrent UTIs, that is three ore more episodes during the preceding 12 months. Suitable patients were randomly assigned to antibiotic treatment with trimethoprim/sulfamethoxazole or to a regimen of oral D Mannose for 24 weeks, and received the other intervention in the second phase of the study.

Outcome measurements and statistical analysis- The time to recurrence of UTI, bladder pain (VAS p) and urinary urgency (VAS u) were evaluated at the end of antibiotic therapy and at the and of 24 weeks fo D Mannose. The results for quantitative variables were expressed as mean values and SD as they were all normally distributed (Shapiro-Wilk test). T-test for paired data was used to analyze differences of time of recurrence, VAS pain, Vas urgency and number of voidings between treatment. Data analysis was performed with STATA statistical package (release 11,1, 2010, Stata Corporation, College Station, Texas, USA).

DETAILED DESCRIPTION:
INTRODUCTION Urinary tract infections (UTIs) are among the most common infectious diseases, with a substantial financial burden to society. In Europe data on the presence of various types of UTIs indicate a high impact on quality of life of people affected, it is important the impact of urinary tract infections on the economy in general and on the health system in particular. In the U.S. urinary tract infections account for more than 7 million doctor visits each year, including more than 2 million visits for cystitis. The bacterium E. coli, which is the source of 90% of urinary tract infections, shows an incredible ability to survive in the human body, and is able to change rapidly to survive antibiotics. An infection of the urinary tract must be stopped before it begins to migrate to the kidneys, where it can cause serious infections. Women with frequent reinfections have a rate of 0.13 to 0.22 UTIs per month (1.6 to 2.6 infections per year). For premenopausal, healthy, and active females, recurrent UTIs are a major healthcare concern. Recurrent urinary tract infection (RUTI) is defined as three episodes of urinary tract infection (UTI) with 3 positive urine cultures in the previous 12 months or two episodes in the last six months. The usual present strategies employing a prophylactic antibiotic regime to prevent recurrent UTIs include long-term low-dose prophylactic antimicrobial treatment or postcoital antibiotic treatment. However, it seems that these strategies do not alter the long-term risk of recurrence. Patients with frequent UTIs who take prophylactic antimicrobial agents for extended periods decrease their infections during prophylaxis, but the rate of infection returns to pre-treatment rates when prophylaxis is stopped . Long-term antibiotics do not appear to positively affect the patient's basic susceptibility to infections. The cell wall of E. coli bacteria has tiny finger-like projections that contain complex molecules called lectins on their surface. These lectins act as a cellular glue that binds the bacteria to the bladder wall so they cannot be easily rinsed out by urination . In this pilot study the aim was to evaluate if oral D Mannose could be used as a safe and effective treatment and as a prophylactic measure for recurrent UTIs in adult women.

PATIENTS AND METHODS Suitable female patients with recurrent urinary tract infections who were visited at the outpatient Clinic of our Urology Department were eligible for study. The work has been conducted in accordance with the principles of the Declaration of Helsinki of World Medical Association. Patients were enrolled in the study after treatment for the most recent urinary tract infection if they had positive urinary cultures at that time.

Each participant entering the trial was assigned to one of the following treatments in a random sequence:

1. A regimen of five-day antibiotic therapy with trimethoprim/sulfamethoxazole 160 mg/800 mg twice a day. Then 1 week of antibiotic every 4 weeks for the following 23 weeks
2. A regimen of oral D Mannose 1 gr. 3 times a day, every 8 hours for 2 weeks, and subsequently 1 gr. twice a day for 22 weeks. D-Mannose has the best activity when urine has neutral pH, therefore patients were instructed to measure urinary pH using dipsticks and use oral sodium bicarbonate 250 mg b.i.d.or potassium citrate 1 gr. b.i.d. as alkalinizing agents if pH was <7.

Patients were randomly assigned to antibiotic treatment with trimethoprim/sulfamethoxazole or to a regimen of oral D Mannose for 24 weeks, and received the other intervention in the second phase of the study.

VAS score for bladder pain (VASp) and for urgency (VASu) was evaluated before starting D Mannose and at 24 weeks. The 24 hour number of voidings was obtained filling a voiding diary before and at the end of treatment with D Mannose. Cure was defined as the resolution of symptoms and no post-treatment bacteriuria at the 24 week follow-up visit. Cure with recurrence was defined as having resolution of symptoms with negative cultures at 12 week followed by significant UTI with bacteriuria before 24 weeks. Failure was defined as having persistent symptoms and significant bacteriuria before 24 weeks. The cure rate was determined for patients who met infection criteria, returned for the follow-up visits and had been treated with an antimicrobial for recurrent urinary tract infection occurring twice or more times during the 6 months preceding the 24 weeks course of daily oral D Mannose. The time to recurrence of UTI, VAS pain and VAS urgency were evaluated at the end of antibiotic therapy and at the end of 24 week treatment with oral D Mannose. Statistical Analysis- The results for quantitative variables were expressed as mean values and SD as they were all normally distributed (Shapiro-Wilk test). T-test for paired data was used to analyze differences of time of recurrence, VAS pain, Vas urgency and number of voidings between treatment. Data analysis was performed with STATA statistical package (release 11,1, 2010, Stata Corporation, College Station, Texas, USA).

DISCUSSION- The approach in the management of recurrent urinary tract infections is usually to treat adequately an episode of infection and after the completion should document complete eradication with a urine culture; if infection reoccurs or persists then imaging is required. In the management of recurrent UTIs in women it is a common practice to fight the resistance of the bacterium E. coli by varying the type of antibiotics, or increasing the dose and duration of therapy. However, in doing so the bacteria become even more resistant to broad spectrum antibiotics. Moreover, the resistance of the bacterium would not increase if the infection was due to a new E. coli contamination of the faeces or to sexual contact. What actually appears to occur is the survival of a part of the old colony of bacteria in the urinary tract, they remain latent and are reactivated by various favourable conditions, the relentless recurrences are therefore not considered as reinfection. It could be learnt a lot from patients and from research done on the causes of repeated urinary tract infections, especially due to the bacterium E. coli. Uropathogenic Escherichia coli (UPEC) strains may contain virulence factors that allow the bacteria to penetrate into the transitional cells and form quiescent intracellular reservoirs (QIRs). Establishment of QIRs throughout the underlying transitional epithelium may predispose an individual to an increased likelihood of recurrence and may account for some of the frequent same-strain recurrences that are seen clinically despite appropriate antibiotic therapy. A difficult aspect of treating urinary tract infections in women is the high likelihood of recurrence. In a series of trials a group of susceptible women averaged 2.6 infections per patient per year despite the apparent effectiveness of short-term therapy. While long-term prophylaxis was relatively effective in that series, resistance to trimethoprim-sulfamethoxazole by urinary pathogens increased to 19% in a 5-year period. Although there is debate regarding the duration of antibiotic therapy, emergence of drug-resistant organisms has to be considered with prolonged antibiotic use, even in healthy women with uncomplicated UTIs. A number of triggers lead to the reactivation of dormant E.coli already in the bladder, or the release of E.coli pods from behind biofilms in the bladder. When a first UTI is caused by E. coli, the risk of a second infection within 6 months is greater than when a first infection is cause by another uropathogen. Although E. coli was the most frequently isolated microorganism in our group of patients, the limited number of patients studied could not confirm this assumption. The chemical structure of D-Mannose causes it to stick to E. coli bacteria, maybe even more tenaciously than E. coli adheres to human cells. Although the mechanism of how it works is complicated, theoretically, if enough D-mannose is present in the urine, it binds to the bacteria and prevents them from attaching to the urinary tract lining. Our clinical experience shows that D Mannose represents a useful choice to address the problem of recurrent UTIs. The time required to develop a new infection, or for the re-emergence of the bacterial reservoir, as can be assumed from new data, is significantly longer with a prolonged course of oral D Mannose than with antibiotic treatment, even when these are used for long periods at a low dose, or in cycles. We actually know mannose has no bactericidal properties, and it might well be that the dosage and duration of therapy have to be individualized according to bacterial growth and replication speed in the bladder and urinary tract. The major part of mannose ingested is eliminated with urine and works by binding to bacteria concentrated in infected urine and attempting to perpetuate infection by binding to mannose receptors of urothelial bladder cells, this mechanism being the one involved in most cases of recurrences. In most cases recurrences are wrongly regarded as re-infections: it is highly likely that bactericidal molecules not possessing the same properties cannot produce the same consistent effect, that is the elimination of more and more loads of bacteria with urine, "alive" albeit inactivated, motionless, devoid of pathogenic potential due to mannose linked to them.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* 3 or more culture documented urinary tract infections in the preceding 12 months
* Patients who had not taken antimicrobials within 4 weeks and were not pregnant or contemplating pregnancy.

Exclusion Criteria:

* Patients with evidence of upper urinary tract infection, such as temperature higher than 38 °C, flank/lumbar pain or tenderness.

Ages: 22 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Porru, MD, Principal Investigator — Urology Dept. Fondazione IRCCS Policlinico San Matteo Pavia
Locations (1):
- Urology Department Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Background] Mulvey MA, Lopez-Boado YS, Wilson CL, Roth R, Parks WC, Heuser J, Hultgren SJ. Induction and evasion of host defenses by type 1-piliated uropathogenic Escherichia coli. Science. 1998 Nov 20;282(5393):1494-7. doi: 10.1126/science.282.5393.1494. PMID 9822381
- [Background] Mulvey MA, Schilling JD, Hultgren SJ. Establishment of a persistent Escherichia coli reservoir during the acute phase of a bladder infection. Infect Immun. 2001 Jul;69(7):4572-9. doi: 10.1128/IAI.69.7.4572-4579.2001. PMID 11402001
- [Background] Mulvey MA, Schilling JD, Martinez JJ, Hultgren SJ. Bad bugs and beleaguered bladders: interplay between uropathogenic Escherichia coli and innate host defenses. Proc Natl Acad Sci U S A. 2000 Aug 1;97(16):8829-35. doi: 10.1073/pnas.97.16.8829. PMID 10922042
- [Derived] Cooper TE, Teng C, Howell M, Teixeira-Pinto A, Jaure A, Wong G. D-mannose for preventing and treating urinary tract infections. Cochrane Database Syst Rev. 2022 Aug 30;8(8):CD013608. doi: 10.1002/14651858.CD013608.pub2. PMID 36041061
- See also: related reference — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC34019/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 female patients aged between 22 and 74 years were visited at the outpatient Clinic (July 2011-July 2012), they were eligible for study if they were 18 years old or older and had 3 or more culture documented urinary tract infections (UTI) in the preceding 12 months. Women were excluded from study if they had evidence of upper UTI
Pre-assignment Details: All patients before entering the trial were prescribed and followed a regimen of continuous, low-dose daily antibiotic prophylaxis at bedtime or post-coital prophylaxis with cotrimoxazole or ciprofloxacin, whenever the UTI occurred 24-48 hours after intercourse.
Groups:
- D Mannose First, Then Trimethoprim/Sulfamethoxazole: D Mannose 1 gr. every 8 hours for 2 weeks, subsequently 1 gr. every 12 hours for 22 weeks then Antibiotic : trimethoprim/sulfametoxazole 80 mg + 400 mg twice a day; length of treatment: 5-7 days
- Trimethoprim/Sulfamethoxazole First, Then D Mannose: Antibiotic : trimethoprim/sulfametoxazole 80 mg + 400 mg twice a day; length of treatment: 5-7 days then D Mannose 1 gr. every 8 hours for 2 weeks, subsequently 1 gr. every 12 hours for 22 weeks
Period: Overall Study
Arm/Group | D Mannose First, Then Trimethoprim/Sulfamethoxazole | Trimethoprim/Sulfamethoxazole First, Then D Mannose
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participamts: D Mannose 1 gr. every 8 hours for 2 weeks, subsequently 1 gr. every 12 hours for 22 weeks then Antibiotic : trimethoprim/sulfamethoxazole 160/800 mg; length of treatment: 5-7 days
Arm/Group | All Study Participamts
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Region of Enrollment [Number; unit: participants]
  Italy | 60
urinary tract infection [Number; unit: participants]
  <18 years | 0
  Between 18 and 74 years | 60
  >75 years | 0
positive urine culture [Number; unit: participants] | 60

OUTCOME MEASURES:

1. Primary Outcome: Days
Description: time required to develop the next urinary tract infection; evaluation by means of urine analysis and urine culture
Time Frame: 168
Measure: Mean (Standard Deviation); unit: days
Groups:
- D Mannose First, Then Trimethoprim /Sulfamethoxazole: 1 gr. every 8 hours for 2 weeks, subsequently 1 gr. every 12 hours for 22 weeks then Antibiotic : trimethoprim/sulfamethoxazole 160/800 mg; length of treatment: 5-7 days
- Trimethoprim /Sulfamethoxazole First, Then D Mannose: trimethoprim/sulfametossazole 160/800 mg for 5-7 days then D Mannose 1 gr. every 8 hours for 2 weeks
Arm/Group | D Mannose First, Then Trimethoprim /Sulfamethoxazole | Trimethoprim /Sulfamethoxazole First, Then D Mannose
Number analyzed (Participants) | 30 | 30
days | 200 (50.7) | 52.7 (11.2)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- D Mannose Versus Antibiotic: 1 gr. every 8 hours for 2 weeks, subsequently 1 gr. every 12 hours for 22 weeks
  D Mannose : D Mannose versus oral antibiotic
  Antibiotic : length of treatment: 5-7 days
Arm/Group | D Mannose Versus Antibiotic
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No